CLINICAL TRIAL: NCT04644055
Title: Endoscopic Ultrasound Share-wave for the Evaluation of Patients With Chronic Liver Disease
Brief Title: EUS Share-wave in Patients With Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: IECED-110520
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Liver Cirrhosis
Keywords: liver cirrhosis; fibrosis; endoscopic ultrasonography; elasticity imaging, tissue
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — EUS-guided liver biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic liver disease with liver cirrhosis: Evaluation of the right and left hepatic lobe with EUS-guided share wave evaluation. All patients with chronic liver disease will have a transient elastography evaluation, EUS- elastography of the liver and an EUS-guided liver biopsy.
  Interventions: Diagnostic Test: EUS- share wave of the liver
- Control patients: Patients without history of chronic liver disease after clinical and transient elastography evaluation will be submitted for EUS-guided share wave evaluation of the liver. Patients were originally undergoing EUS evaluation for evaluation of suspected subepithelial lesions.
  Interventions: Diagnostic Test: EUS- share wave of the liver

INTERVENTIONS:
Diagnostic Test: EUS- share wave of the liver — Evaluation of the right and left hepatic lobe with EUS-guided share wave

SUMMARY:
Patients with chronic liver disease may develop progressive hepatic fibrosis. Liver cirrhosis should be detected at the early stages in order to avoid the complications related to these two conditions.

The diagnostic work-up of patients with chronic liver disease includes less-invasive diagnostic methods such as abdominal ultrasonography, transient elastography, upper endoscopy; and more invasive procedures, mainly liver biopsy and portal pressure gradient measurement, both with associated risks.

Endoscopic ultrasound offers a benefit of including all diagnostic work-up in a single procedure. The investigators previously demonstrated that EUS-elastography of the liver and spleen is reliable marker for predicting liver cirrhosis.

Recently, a quantitative evaluation of fibrosis using share wave elastography was introduced, mainly for the pancreatic tumor fibrosis measurement (2). Elastography measures the elasticity of tissues (hardness); whereas share wave measures the tissue elasticity as the elastic modulus by measuring the share wave velocity. Share wave measurement will be performed with the Arietta 850 Endoscopic ultrasound console using a linear ultrasound video gastroscope EUS-J10 (Pentax Medical, Hoya Corp, Japan). The investigators proposed the EUS-share wave of the liver as a reliable diagnostic marker in patients with liver cirrhosis.

DETAILED DESCRIPTION:
A non-blinded, prospective trial. Primary disease condition: liver cirrhosis Keywords: Liver Cirrhosis; Fibrosis; Endoscopic Ultrasonography; Elasticity Imaging, Tissue.

Study Design: Observational study model: a non-blinded, non-randomized, prospective trial Time perspective: prospective Enrollment type: actual Number of subjects: 16 participants Number of groups/cohorts: 2 cohorts Target follow-up duration: 6 months

Based on the proportion of patients with the liver strain histogram (LSH) >87.40 among cirrhosis (87.5%) and control cases (31.0%) described by Robles-Medranda et al. (1), the investigators calculated eight patients per study group with a 5% and 20% of alpha and beta error respectively, with an 80% of power statistic.

ELIGIBILITY:
Inclusion Criteria:

* Provided informed written consent
* Age greater than 18 years of age
* Confirmed diagnosis of chronic liver disease based on transient elastography
* Patients with EUS-guided liver biopsy

Exclusion Criteria:

* History of uncontrolled coagulopathy
* Contraindications to EUS-guided liver biopsy
* Pregnancy or nursing
* History of hepatocellular carcinoma
* Patients with equivocal transient elastography results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Performed at Instituto Ecuatoriano de Enfermedades Digestivas (IECED), an academic tertiary center in Guayaquil, Ecuador. Patients will be invited to participate during outpatient clinic visits.
  All consecutive participants need to be ≥18 years old and has a history of chronic liver disease with histological proven liver cirrhosis. Control patients will be patients without history of chronic liver disease and will be included following a transient elastography test within normal limits.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Correlation of EUS-share of the liver | 2 months
  Evaluation of the correlation between transient elastography, EUS-elastography of the liver, EUS-guided liver biopsy and EUS-guided share wave of the liver
Diagnostic accuracy of EUS-share wave of the liver | 2 months
  Evaluate the diagnostic accuracy of EUS- share wave of the liver for predicting liver cirrhosis. Receiver operating characteristic curve development with evaluation of the sensitivity, specificity, PPV and NPV of EUS-guided share wave of the liver to predict liver cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, MD FASGE, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Robles-Medranda C, Oleas R, Puga-Tejada M, Valero M, Valle RD, Ospina J, Pitanga-Lukashok H. Results of liver and spleen endoscopic ultrasonographic elastography predict portal hypertension secondary to chronic liver disease. Endosc Int Open. 2020 Nov;8(11):E1623-E1632. doi: 10.1055/a-1233-1934. Epub 2020 Oct 22. PMID 33140018